CLINICAL TRIAL: NCT02301182
Title: A Single-Center Randomized, Patient-Blinded, Prospective Five-Year Study to Compare the Functional Results After Insertion of ADM X3-MoP Cup (Stryker) and a CoC Cup (Zimmer) in Primary THA
Brief Title: Comparison of Functional Results of ADM X3-MoP Cup (Stryker) and a CoC Cup (Zimmer) in Young Patients
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: VEK-44819
Record Dates: First submitted 2014-10-21; First posted 2014-11-25 (Estimated); Last update posted 2024-01-11 (Actual); Status verified 2024-01

CONDITIONS: Arthroplasties, Hip Replacement

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- ADM X3-MoP Cup (Active Comparator): THA: ADM dual-mobility hydroxyapatite coated cups with X3TM HXLPE liners on 28mm BIOLOX® delta femoral heads (Stryker) with femoral stems being 2nd generation Accolade stems of the taper lock type, proximal circumferential coated with a 50µm plasma-spray PureFix HA coating to aid the mechanical engagement in bone coating (Stryker)
  Interventions: Device: ADM X3-MoP Cup
- CoC Cup (Active Comparator): THA: CoC BIOLOX® delta-delta large-head single-mobility cementless fiber-mesh titanium coated acetabular system from Zimmer (Zimmer TrilogyIT cup/CLS spotorno stem) with a grit-blasted osteophilic titanium alloy CLS® Spotorno femoral stems (Zimmer) that has a three-dimensional wedge shape and sharpened ribs in the proximal region
  Interventions: Device: CoC Cup

INTERVENTIONS:
Device: ADM X3-MoP Cup
  Arms: ADM X3-MoP Cup
Device: CoC Cup
  Arms: CoC Cup

SUMMARY:
A Single-Center Randomized, Patient-Blinded, Prospective Five-Year Study to Compare the Functional Results after Insertion of ADM X3-MoP Cup (Stryker) and a CoC Cup (Zimmer) in Primary THA. 60 patients will be enrolled during a 2 year period. At surgery tantalum beads will be inserted into predrilled holes of the polyethylene rim for assessment of motion of the large mobile poly in the ADM Trident Cup by use of RSA. Patients will be followed by functional examinations as well as PROM assessment.

DETAILED DESCRIPTION:
With Metal-on-Metal (MoM) articulations leaving the marked the THA bearing choice for younger patients is currently debated and overall the choice stands between CoC and MoP. New HXLPE is wear-resistant and safe and clinical HXLPE wear (RSA) hardly exceed the wear measured in retrieval CoC implants. For CoC articulations stripe wear on edge loading is a reported problem leading to increased wear in examined retrieval components and CoC wear is dependent on component position. Although the risk is very small, CoC bearings are at still at risk of fracture, and functional squeaking is a complication that adversely affects the quality of life in about 1% of CoC THA patient. Dual mobility MoP cups were designed for reducing hip dislocations in older patients treated with THA after medial hip fractures. The concept provides good stability and mobility and may also be an optimal solution for younger and active patients; however, dual mobility MoP has not previously been documented for use in younger patients. The anatomical dual mobility (ADM) cup design (Stryker) is soft tissue sparing (iliopsoas tendon) potentially leading to lesser groin-pain and squeaking is not a concern. It is currently unknown if the outer-articulation of the dual mobility PE liner keeps moving over time or could impinge in the joint capsule in an undesirable position and result in unwanted edge loading and higher wear-rates. Metal ions are produced even in MoP bearings and even though in dual-articulation MoP bearings most (90%) of the motion is believed to occur between the head and liner (ceramic-polyenthylene), the metal ion levels may be higher than expected for MoP hips (large poly contact in metal shell), while expectedly there will be no metal ions in CoC THA.

ELIGIBILITY:
Inclusion Criteria:

* primary hip osteoarthritis
* sufficient bone quality for total hip arthroplasty
* age 40 through 65 years of age
* informed and written consent
* patient can only enter the project with one hip

Exclusion Criteria:

* neuromuscular or vascular disease in the affected leg
* patients with osteoporosis
* fracture sequelae or previous extensive hip surgery
* patients with metabolic bone disease including rheumatoid arthritis
* non-Danish citizenship
* patients who do not comprehend the Danish language
* senile dementia
* alcoholism and drug abuse
* major psychiatric disease
* current metastatic cancer disease and on-going treatment with radiation therapy/chemotherapy
* severe systemic disease affecting gait
* contralateral knee, hip and/or spine disease
* on-going case regarding industrial injury insurance of the hip
* patients with very poor dental status

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2014-11; Primary Completion 2026-06 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
Motion analysis (accelerometer (Ax3 Axivity) based activity monitoring) | 5 year
  For all participants: Inertia sensors are a new technology for patient motion analysis which allows simple and fast routine clinical movement analysis and long-term activity monitoring. We will employ the newest generation of accelerometer (Ax3 Axivity) based activity monitoring (small, light, low cost, validated for orthopaedic patients also with walking aids) to count, in real life, the number of events and the duration of postures and activities. Further muscle power investigations such as by use of the legg extension power rig will be used.
questionnaires ("the Harris Hip Score" (HHS), the Oxford Hip Score (OHS), the HOOS score, satisfaction, dislocation, and revisions) | 5 year
  For all participants: Pre- and postoperative clinical evaluations will be made according to "the Harris Hip Score" (HHS), the Oxford Hip Score (OHS), the HOOS score, and satisfaction, dislocations and revisions will be noted. Moreover, pre-operative rest and motion pains will be assessed by visual analogue scale scores (VAS).
Radiography (implant migration and wear) | 5 year
  For all participants: Within a week following surgery a stereo x-ray is performed and this functions as the baseline for future follow-up (in this study at 1 year, 2 years and 5 years). When comparing all stereo x-rays in a patient series, implant migration with respect to a set of bone markers can be calculated in three dimensions as a function of time - similarly wear of the implant surfaces can be evaluated.Fluoroscopic stereoradiometric recordings (Dynamic RSA) can be used to assess the functional motion of implants at desired motion speeds. In this study we record the liner motion of the ADM cup with the patients in different positions that in theory stresses the motion of the liner into new positions at edge-motions. The purpose is to gain knowledge on the safety function of the implant in vivo - if the liner moves and if it positions safely like it is supposed to.

CONTACTS AND LOCATIONS:
Locations (1):
- Aarhus University Hospital, Aarhus, Denmark

REFERENCES:
- [Derived] Jorgensen PB, Kaptein BL, Soballe K, Jakobsen SS, Stilling M. Combined and hybrid marker models for radiostereometry assessment of polyethylene liner motion in dual mobility hip prosthesis: a proof-of-concept study. Eur Radiol Exp. 2021 Dec 15;5(1):55. doi: 10.1186/s41747-021-00253-x. PMID 34907467